CLINICAL TRIAL: NCT01690975
Title: A Phase I, Randomized, Placebo-controlled, Dose Escalation Study to Assess the Tolerability of Benzonatate Following Single Dose Administration in Healthy Volunteers
Brief Title: Benzonatate Dose Tolerance Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B3551001; BT-10-29
Record Dates: First submitted 2012-07-05; First posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — benzonatate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo Control
  Interventions: Drug: Placebo
- Benzonatate (Experimental): Benzonatate Active
  Interventions: Drug: Benzonatate - 400 mg; Drug: Benzonatate - 600 mg

INTERVENTIONS:
Drug: Placebo — Placebo - single dose at start of each treatment period
  Arms: Placebo
Drug: Benzonatate - 400 mg — Benzonatate - 400 mg single dose
  Arms: Benzonatate
Drug: Benzonatate - 600 mg — Benzonatate - 600 mg single dose
  Arms: Benzonatate

SUMMARY:
This is a single-center, randomized, third party blind, placebo controlled, dose escalation study of benzonatate following single dose administration. The primary oobjective is to assess the safety and tolerability of increasing oral doses of benzonatate following single dose administration in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG, or clinical laboratory tests.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results, and in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose
Plasma Decay Half-Life (t1/2) | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD): Assessed at end of study | End of study (2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3551001&StudyName=Benzonatate%20Dose%20Tolerance%20Study